CLINICAL TRIAL: NCT03371238
Title: The Effect of Floorball on Health and Performance Parameters in Healthy Seniors
Brief Title: Effect of Floorball on Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, PhD, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MFloorball
Record Dates: First submitted 2017-11-17; First posted 2017-12-13 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Aging Problems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Floorball (Experimental)
  Interventions: Behavioral: Floorball
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Floorball — The subjects in this group are set to play floorball three times pr. week for 39 weeks.
  Arms: Floorball

SUMMARY:
To investigate the effect of floorball on health and performance in healthy subjects over 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* age 65-85
* physical activity <2 hours pr. week.

Exclusion Criteria:

* age <18 years
* Injuries that prevent the subject from playing floorball
* Alcohol >14 units pr. week.
* Pregnancy
* Other serious conditions

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Echocardiogram | Changes from baseline measured after 12 weeks and 39 weeks
  The measure of the hearts geometric dimensions
Bodycomposition | Changes from baseline measured after 12 weeks and 39 weeks
  DXA scan

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark